CLINICAL TRIAL: NCT02318407
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AMG 403 in Younger and Older Subjects With Osteoarthritis Knee Pain
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AMG 403 in Subjects With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060145
Record Dates: First submitted 2014-12-02; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — AMG 403

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 403 (Experimental): AMG 403 administered as subcutaneous doses
  Interventions: Drug: AMG 403
- Placebo (Placebo Comparator): No active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 403 — AMG 403 for the treatment of subjects with osteoarthritis
  Arms: AMG 403
Drug: Placebo — contains no active drug
  Arms: Placebo

SUMMARY:
This is a sequential, randomized, double-blind, placebo controlled, multiple dose, dose escalation study in subjects with OA knee pain (n=32; 8/cohort). In each cohort, subjects will be randomized 3:1 to receive SC AMG 403 or placebo once every 4 weeks for a total of 4 doses (Q28D x 4).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA as determined by ACR criteria: Knee pain and radiographic osteophytes and at least 1 of the following 2 items: Morning stiffness 30 minutes, Crepitus on motion, a VAS pain score of ≥ 30 mm for index knee at screening,

Exclusion Criteria:

* Weight of > 125 kg, Inflammatory arthropathy including secondary OA (eg, degenerative arthritis in patients with rheumatoid arthritis) as confirmed by a rheumatologist or investigator, Diagnosis of a condition other than knee OA that, in the investigator's opinion, may cause or affect pain or pain assessment in the index knee; these conditions may include but are not limited to radiculopathy or neuropathy, vasculopathy, fibromyalgia or active depression, Subjects taking neuromodulatory agents (antiepileptics or antidepressants) used as analgesic therapy for neuropathic pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by subject incident of treatment-emergent adverse events, clinically significant changes in vital signs, physical examinations endpoints, clinical laboratory safety tests, and ECGs | from 197 days to 211 days
  Subject incident of treatment-emergent adverse events, clinically significant changes in vital signs, physical examinations endpoints, clinical laboratory safety tests, and ECGs

SECONDARY OUTCOMES:
Pharmacokinetics profile of AMG 403 including Tmax, AUClast and Cmax | from 197 days to 211 days
  serum concentrations and derived PK parameters of AMG 403

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Gow JM, Tsuji WH, Williams GJ, Mytych D, Sciberras D, Searle SL, Mant T, Gibbs JP. Safety, tolerability, pharmacokinetics, and efficacy of AMG 403, a human anti-nerve growth factor monoclonal antibody, in two phase I studies with healthy volunteers and knee osteoarthritis subjects. Arthritis Res Ther. 2015 Oct 8;17:282. doi: 10.1186/s13075-015-0797-9. PMID 26449617
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com